CLINICAL TRIAL: NCT04212793
Title: Detection of Pituitary Neuroendocrine Tumor (PitNET) Tissue During Endoscopic Transsphenoidal Surgery Using Bevacizumab-800CW
Brief Title: Detection of PitNET Tissue During TSS Using Bevacizumab-800CW
Acronym: DEPARTURE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Jos M. A. Kuijlen, Principal Investigator, University Medical Center Groningen
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: UMCG 201800170
Record Dates: First submitted 2019-12-17; First posted 2019-12-30 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Pituitary Tumor; Pituitary Adenoma; Pituitary Macroadenoma
MeSH Terms: conditions — Pituitary Neoplasms

STUDY DESIGN:
Intervention Model Description: The study is a non-randomized, non-blinded, prospective, single center, pilot dose-finding study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- NIR endoscopic TSS with 4.5 mg bevacizumab-800CW (Experimental): IV-administration of 4.5 mg of the fluorescent tracer bevacizumab-800CW to 3 patients with a pituitary neuroendocrine tumor (PitNET) with a Knosp grade of 3 or 4. The optimal dose will be expanded to include 6 patients.
  Interventions: Drug: Bevacizumab-IRDye800CW; Device: Molecular Fluorescence Endoscopy platform
- NIR endoscopic TSS with 10 mg bevacizumab-800CW (Experimental): IV-administration of 10 mg of the fluorescent tracer bevacizumab-800CW to 3 patients with a pituitary neuroendocrine tumor (PitNET) with a Knosp grade of 3 or 4. The optimal dose will be expanded to include 6 patients.
  Interventions: Drug: Bevacizumab-IRDye800CW; Device: Molecular Fluorescence Endoscopy platform
- NIR endoscopic TSS with 25 mg bevacizumab-800CW (Experimental): IV-administration of 25 mg of the fluorescent tracer bevacizumab-800CW to 3 patients with a pituitary neuroendocrine tumor (PitNET) with a Knosp grade of 3 or 4. The optimal dose will be expanded to include 6 patients.
  Interventions: Drug: Bevacizumab-IRDye800CW; Device: Molecular Fluorescence Endoscopy platform

INTERVENTIONS:
Drug: Bevacizumab-IRDye800CW — Intravenous administration of 4.5, 10 or 25 mg of Bevacizumab-IRDye800CW prior to endoscopic transsphenoidal surgery
  Other Names: Tracer administration
Device: Molecular Fluorescence Endoscopy platform — A flexible fluorescence fiber-bundle is attached to a fluorescence camera platform to enable the detection of fluorescence signals. The fluorescence fiber-probe is inserted through the standard working channel of the Surgvision explorer endoscope. During surgery, three imaging moments are defined in which the fluorescence molecular endoscopy system will detect the fluorescent signal
  Other Names: Fluorescence endoscopy

SUMMARY:
There is a need for improved visualization of presence and extent of pituitary neuroendocrine tumor (PitNET) tissue during transsphenoidal surgery (TSS), especially in tumors invading the cavernous sinus (CS). Optical molecular imaging of PitNET associated biomarkers is a promising technique to accommodate this need. Vascular Endothelial Growth Factor (VEGF-A) is overexpressed in PitNET tissue compared to normal pituitary tissue and has proven to be a valid target for molecular imaging. Bevacizumab is an antibody that binds VEGF-A. By conjugating a fluorescent dye to this antibody, the fluorescent tracer molecule bevacizumab-800CW is created, which binds to VEGF-A. The investigators hypothesize that bevacizumab-800CW accumulates in PitNET tissue, enabling visualization using a molecular fluorescence endoscopy system. In this pilot intervention study the investigators will determine the feasibility of using microdoses (4.5, 10 and 25 mg) of bevacizumab-800CW to detect PitNET tissue intraoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an established diagnosis of PitNET with a Knosp grade of 3 or 4 who are scheduled to undergo TSS.
* WHO performance status 0-2
* Signed written informed consent

Exclusion Criteria:

* Medical or psychiatric conditions that compromise the patient's ability to give informed consent
* Pregnant or lactating women. Documentation of a negative pregnancy test must be available for woman of childbearing potential. Woman of childbearing potential are pre- menopausal women with intact reproductive organs and women less than two years after menopause
* History of infusion reactions to bevacizumab or other monoclonal antibody therapies.
* Inadequately controlled hypertension with or without current antihypertensive medication
* Within 6 months prior to inclusion: myocardial infarction, TIA, CVA, pulmonary embolism, uncontrolled chronic hepatic failure, unstable angina pectoris

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-10-28 (Actual); Primary Completion 2022-10-24 (Actual); Study Completion 2022-10-24 (Actual)

PRIMARY OUTCOMES:
Discrimination of tumorous and non-tumorous tissue based on in vivo and ex vivo fluorescence measurements from bevacizumab-800CW gained during fluorescence endoscopic transsphenoidal surgery of pituitary neuroendocrine tumors (PitNETs) | Three days after tracer injection
  To determine the sensitivity of the marker bevacizumab-800CW in discriminating between tumorous and non-tumorous tissue during endoscopic transsphenoidal surgery of pituitary neuroendocrine tumors (PitNETs) defined as the tumor to background ratio and intrinsic fluorescence
Number of participants with adverse events (AE), serious adverse events (SAE) and suspected unexpected serious adverse reactions (SUSAR) | Up to 7 days after tracer injection
  Data collection as a measure of safety and tolerability regarding administration of bevacizumab-800CW

SECONDARY OUTCOMES:
The correlation of in vivo and ex vivo fluorescent signals to histopathological analysis results | Up to 1,5 year
  Correlate the H/E images to the fluorescent images made with multiple ex vivo imaging modalities
Quantification of the fluorescent signal by MDSFR/SFF spectroscopy | Up to 1,5 year
  Multi-diameter single-fiber reflectance with single-fiber fluorescence (MDSFR/SFF) spectroscopy can measure the fluorescence signal quantitatively, both in vivo and ex vivo
Assessment of the (sub)-cellular distribution of bevacizumab-800CW by ex vivo fluorescence microscopy | Up to 1,5 year
  Imaging of the distribution of bevacizumab-800CW with a fluorescence microscope

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schmidt I, Vergeer RA, Postma MR, van den Berg G, Sterkenburg AJ, Korsten-Meijer AGW, Feijen RA, Kruijff S, van Beek AP, den Dunnen WFA, Robinson DJ, van Dijk JMC, Nagengast WB, Kuijlen JMA. Fluorescence detection of pituitary neuroendocrine tumour during endoscopic transsphenoidal surgery using bevacizumab-800CW: a non-randomised, non-blinded, single centre feasibility and dose finding trial [DEPARTURE trial]. Eur J Nucl Med Mol Imaging. 2025 Jan;52(2):660-668. doi: 10.1007/s00259-024-06947-9. Epub 2024 Oct 11. PMID 39390132
- [Derived] Vergeer RA, Postma MR, Schmidt I, Korsten-Meijer AG, Feijen RA, Kruijff S, Nagengast WB, van Dijk JMC, den Dunnen WFA, van Beek AP, Kuijlen JMA, van den Berg G. Detection by fluorescence of pituitary neuroendocrine tumour (PitNET) tissue during endoscopic transsphenoidal surgery using bevacizumab-800CW (DEPARTURE trial): study protocol for a non-randomised, non-blinded, single centre, feasibility and dose-finding trial. BMJ Open. 2021 Oct 7;11(10):e049109. doi: 10.1136/bmjopen-2021-049109. PMID 34620658